CLINICAL TRIAL: NCT03990285
Title: Multimodality 18F-Fluciclovine PET, MRI and Cell Free Circulating DNA to Differentiate Tumor Progression From Pseudoprogression in Patients With Glioblastoma
Brief Title: [18F]Fluciclovine in Post-treatment Glioblastoma ( Axumin )
Acronym: Axumin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ali Nabavizadeh (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor-Investigator, Ali Nabavizadeh, Principal Investigator, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 08319/ IRB# 832812
Record Dates: First submitted 2019-06-06; First posted 2019-06-18 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Glioma Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: To compare 18F-fluciclovine PET uptake measures in glioblastoma patients with tumor progression vs pseudoprogression. To determine a multidimensional signature using 18F-fluciclovine PET, MRI, and plasma cfDNA that accurately differentiates tumor progression from pseudoprogression in post-chemoradiation GBM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [18F]Fluciclovine in glioblastoma (Other): Axumin is a positron emitting radiopharmaceutical that has been studied in vivo in humans in a number of tumor types with positron emission tomography (PET/CT). 18F-Fluciclovine is a fluorine-18 labeled synthetic amino acid analog that is FDA approved as a PET imaging agent for prostate cancer recurrence, however, it has also been tested in other tumors. Investigators will use a typical dose of 18F-fluciclovine that is used for clinical studies in glioblastoma. This will be 5 mCi (approximate range for most studies is anticipated to be 5 mCi +/- 20%), but a lesser dose may be injected if, in the opinion of a Nuclear Medicine Authorized User, complete imaging data could be generated.
  Interventions: Drug: Axumin, Intravenous Solution

INTERVENTIONS:
Drug: Axumin, Intravenous Solution — To compare 18F-fluciclovine PET uptake measures in glioblastoma patients with tumor progression versus pseudoprogression

SUMMARY:
Subjects with histologically proven glioblastoma (GBM) who are suspected to have progression and are candidates for a surgical resection according to standard of care may be eligible for this study. Subjects may participate in this study if they are at least 18 years of age.

Positron emission tomography (PET/CT) imaging will be used to evaluate fluciclovine uptake at sites of suspected progression before planned surgery. In addition, clinical brain MRI with and without contrast will be used to evaluate the tumor pre-operatively. This is a non-therapeutic trial in that imaging will not be used to direct treatment decisions.

Investigators anticipate enrolling up to 30 subjects who will undergo a clinical brain MRI examination with and without contrast and a research 18F-Fluciclovine PET/CT scan of the brain prior to surgery. They will also have a blood draw preoperatively to collect samples for cfDNA analysis. PET/CT imaging sessions will include an injection of approximately 5 mCi (range for most studies is anticipated to be 5 mCi +/- 20%) of 18F-Fluciclovine.

DETAILED DESCRIPTION:
This is a pilot study in subjects with a histologically proven diagnosis of glioblastoma (GB) who have completed chemoradiation and now have new contrast enhancing lesions or lesions showing increased enhancement ( 25% increase) who are recommended for a clinical surgical resection. Subjects may participate in this study if they are at least 18 years of age, most participants will be receiving care at the clinical practices of the University of Pennsylvania. Subjects who come to the University of Pennsylvania for diagnosis and/or treatment of GB and who meet the study inclusion criteria may be approached by study personnel for recruitment into this study. Subjects will be approached about study participation regardless of race or ethnic background. Investigators anticipate enrolling up to 30 participants. Subjects who consent but do not complete the study imaging will be considered not evaluable and will be replaced. Accrual will likely occur over approximately 1-2 years. After undergoing screening assessments and verifying eligibility for study participation subjects will undergo a research 18FFluciclovine PET/CT scan of the brain and a clinical brain MRI with and without gadolinium contrast, all baseline imaging will be done prior to (within 1 week) of the surgical procedure. The PET-CT and MRI can be performed in any order.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. Initial diagnosis of glioblastoma (histologic or molecular proof)
3. Completion of chemoradiation
4. New contrast-enhancing lesion or lesions showing increased enhancement (>25% increase) on standard MRI after completion of chemoradiation
5. Recommended for clinically surgical resection
6. Life expectancy of greater than 3 months in the opinion of an investigator or treating physician.
7. Karnofsky performance status ≥ 60
8. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures

Exclusion Criteria:

1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
2. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
4. Contraindications to MRI or use of gadolinium contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Pseudoprogression or tumor progression by histopathology | 2Years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125